CLINICAL TRIAL: NCT03970109
Title: Human Laboratory Study of ANS-6637 for Alcohol Use Disorder
Brief Title: HLAB-002 of ANS-6637 for Alcohol Use Disorder
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated early following enrollment of n=43 due to clinically significant increases in liver enzymes in 3 women following at least 3 weeks of dosing with both doses of ANS-6637.
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HLAB-002
Record Dates: First submitted 2019-05-28; First posted 2019-05-31 (Actual); Results first posted 2022-03-10 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Alcohol Use Disorder
Keywords: pharmacotherapy; human laboratory study; novel medication
MeSH Terms: conditions — Alcoholism | interventions — ANS-6637

STUDY DESIGN:
Intervention Model Description: This study is a 3-arm, double-blind, randomized, placebo-controlled, parallel group, 3-site study designed to assess the effects of ANS-6637 as compared with placebo on responses to in vivo alcohol cue exposure in the human laboratory setting.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- ANS-6637 - 200mg (Active Comparator): 200 mg ANS-6637 (given as 2 x 100 mg tablet) once a day
  Interventions: Drug: ANS-6637
- ANS-6637 - 600mg (Active Comparator): 600 mg ANS-6637 (given as 2 x 300 mg tablet) once a day
  Interventions: Drug: ANS-6637
- Matched Placebo (Placebo Comparator): 2 placebo tablets once a day
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: ANS-6637 — 200 mg (given as 2 x 100 mg tablet) and 600 mg (given as 2 x 300 mg tablet) once a day
  Arms: ANS-6637 - 200mg; ANS-6637 - 600mg
Drug: Placebo oral tablet — Placebo oral tablet
  Arms: Matched Placebo

SUMMARY:
Primary: The primary objective of this study was to evaluate the effects of 2 different doses of ANS-6637, 200 mg (given as 2 x 100 mg tablets) and 600 mg (given as 2 x 300 mg tablets) once a day, and matched placebo, on alcohol cue-elicited alcohol craving during a human laboratory paradigm after 1 week of daily dosing among subjects with moderate to severe alcohol use disorder (AUD) as confirmed by the Diagnostic and Statistical Manual of Mental Disorders - Fifth Edition (DSM-5™).

Secondary: Secondary objectives included evaluation of ANS-6637 200 mg, ANS-6637 600 mg, and matched placebo on reduction of alcohol consumption, alcohol craving, cigarette smoking (among smokers) and nicotine use (among nicotine users), mood, sleep, alcohol use negative consequences, study retention, and safety and tolerability throughout the last 4 weeks of the treatment phase of the study.

DETAILED DESCRIPTION:
Methodology: This study was a 3-arm, double-blind, randomized, placebo-controlled, parallel group, 3-site study designed to assess the effects of ANS-6637 as compared with placebo on responses to in vivo alcohol cue exposure in the human laboratory setting. After signing informed consent, subjects were screened for eligibility and had other baseline assessments. Screening was permitted over a 14-day period and most baseline assessments were performed on the day of randomization. If eligible for the study, 81 subjects were to be randomized using a stratified permuted block randomization procedure in an approximate 1:1:1 ratio (targeting 27 subjects per group and 27 subjects per each of 3 clinical sites) to receive either ANS-6637 200 mg once daily, ANS-6637 600 mg once daily, or matched placebo for 5 weeks. Clinical site was used as the stratification variable. Subjects were seen in the clinic at screening, at randomization and 5 other times during the study. A final followup telephone interview was conducted 2 weeks after the end of study in-clinic visit. After the first week of investigational product (IP) administration at Study Week 2, subjects underwent a cue reactivity session including 4 individual visual analog scale (VAS) items assessing alcohol craving and one item assessing beverage liking.

Number of Subjects (planned and analyzed): 81 planned; 43 analyzed. The study was put on clinical hold and then stopped early due to clinically significant AEs.

Investigational Product, Dosage, and Mode of Administration:

The target doses were 200 mg (2 x 100 mg tablets) and 600 mg (2 x 300 mg tablets) of ANS-6637 by oral administration once daily for 5 weeks. Subjects in the placebo group took an equivalent number of identically matched placebo tablets (2 per day) by oral administration once daily for 5 weeks.

Duration of Treatment: Each subject participated in the study for up to 10 weeks, including up to 2 weeks of screening, 5 weeks of treatment, one end-of-study visit during the week following the last treatment dose, and a final telephone contact 2 weeks after completing treatment for a safety follow-up.

Statistical Methods (Data Analysis): The original analytical plan was revised slightly due to early stopping of the study as only approximately half of the subjects were randomized to the study at that time.

Analysis Populations:

Modified intention-to-treat (mITT) Analysis Set: The mITT set was defined as subjects randomized to participate in the study that took at least one dose of IP and had a non-missing VAS craving primary endpoint.

Safety Analysis Set: The safety analysis set includes all subjects who took at least one dose of IP.

As the study closed prematurely, only the mITT and Safety Analysis sets were evaluated.

Analysis of the Primary Efficacy Endpoint: Each mITT subject had an initial alcohol cue for "strength" of alcohol craving score from the VAS that was the primary endpoint. Analysis of covariance (ANCOVA) with the "strength" of alcohol craving value as the dependent variable and the pretreatment "strength' of alcohol craving score from the first alcohol cue were an independent fixed effect. Clinical site was included as an independent factor. There were 3 comparisons (ANS-6637 600 mg vs placebo; ANS-6637 200 mg vs. placebo; and ANS-6637 600 mg vs. ANS-6637 200 mg). The Tukey's method was used to adjust for multiple comparisons. No imputation for missing endpoint data was performed.

Analysis of the Secondary Endpoints: There were 3 additional questions asked during the cue session for each beverage cue. Each of these questions was analyzed in the same manner as the primary endpoint. Continuous secondary endpoints during the last 4 weeks of treatment period were analyzed using a mixed-effects model with site, assessment time, and baseline drinking as fixed factors. Models also included time by treatment group interaction term. Analysis of the dichotomous secondary endpoints during the last 4 weeks of treatment period were conducted via logistic regression. No imputation for missing endpoint data was performed for secondary endpoints.

ELIGIBILITY:
Inclusion criteria:

1. Be at least 21 years of age.
2. Meet the DSM-5 criteria for alcohol use disorder of at least moderate severity.
3. If male, report drinking a weekly average of at least 35 drinks per week or if female report drinking a weekly average of at least 28 drinks per week for the 28-day period prior to consent.
4. Have at least 1 heavy drinking day (4 or more drinks for women/5 or more drinks for men) during the 7-day period prior to randomization.
5. Be seeking treatment for AUD and desire a reduction or cessation of drinking.
6. Be able to verbalize an understanding of the consent form, able to provide written informed consent, verbalize willingness to complete study procedures, able to understand written and oral instructions in English and able to complete the questionnaires required by the protocol.
7. Agree (if the subject is female and of child bearing potential) to use at least one of the following methods of birth control to at least 7 days post the last dose of study drug, unless she is surgically sterile, partner is surgically sterile or she is postmenopausal (one year):

   1. oral contraceptives,
   2. contraceptive sponge,
   3. patch,
   4. double barrier (diaphragm/spermicidal or condom/spermicidal),
   5. intrauterine contraceptive system,
   6. etonogestrel implant,
   7. medroxyprogesterone acetate contraceptive injection,
   8. complete abstinence from sexual intercourse, and/or hormonal vaginal contraceptive ring.
8. Agree (if male) to use acceptable methods of contraception if the male participant's partner could become pregnant from the time of the first administration of the study drug until 7 days following the final administration of the study drug. One of the following acceptable methods of contraception must be utilized:

   1. Surgical sterilization (vasectomy);
   2. The participant's female partner uses oral contraceptives (combination estrogen/progesterone pills), injectable progesterone or sub dermal implants (commenced at least 14 days prior to study drug administration to the male participant)
   3. The participant's female partner uses a medically prescribed topically applied transdermal contraceptive patch (commenced at least 14 days prior to study drug administration to the male participant);
   4. The participant's female partner has undergone tubal ligation (female sterilization) or is postmenopausal (one year);
   5. The participant's female partner has undergone placement of an intrauterine device or intrauterine system;
   6. True abstinence: when this is in line with the preferred and usual lifestyle of the participant.
9. Agree (if male) to refrain from sperm donation from the randomization visit to at least 7 days after the last dose of study drug.
10. Be able to take oral medication and be willing to adhere to the medication regimen.
11. Complete all assessments required at screening and baseline.
12. Have a place to live in the 2 weeks prior to randomization and not be at risk that s/he will lose his/her housing in the next 2 months.
13. Not anticipate any significant problems with transportation arrangements or available time to travel to the study site over the next 2 months.
14. Not have any unresolved legal problems that could jeopardize continuation or completion of the study.
15. Provide contact information of someone, such as a family member, spouse, or significant other, who may be able to contact the subject in case of a missed clinic appointment.
16. Have a BAC by breathalyzer equal to 0.000 when s/he signed the informed consent document.
17. If taking a medication for depression or anxiety, must have been taking a stable dose in the 2-months prior to randomization and plan to continue during the study. This includes drugs such as the following:

    1. Selective serotonin reuptake inhibitors (SSRIs)
    2. Dual uptake inhibitors
    3. Serotonin-norepinephrine reuptake inhibitors (SNRIs)
    4. Tricyclic antidepressants
    5. Monoamine oxidase inhibitors (MAOIs)
18. Be someone who in the opinion of the investigator would be expected to complete the study protocol.
19. Agree to the schedule of visits, verbally acknowledge that s/he will be able to attend each scheduled visit, participate in phone visits and that s/he does not have any already scheduled events or a job that may substantially interfere with study participation.
20. Be willing to use a smartphone's video capability to record daily oral ingestion of tablets for the entire 5-week treatment period (subject's own smartphone or one provided by AiCure).
21. Have sitting (3 to 5 minutes) vital signs at the screening visit within the following limits:

    1. Systolic blood pressure 90 to 160 mmHg
    2. Diastolic blood pressure of 50 to 95 mmHg
    3. Heart rate of 40 to 90 beats per minute Note: Vital signs may be repeated once if outside the limits above and if within the limits on a second evaluation, the subject may be included.

Exclusion Criteria:

1. Current (past 12 months) substance use disorder of at least moderate severity (4 or more criteria) for any psychoactive substance other than alcohol and nicotine, including sedatives and hypnotics, as defined by DSM-5 criteria.
2. Urine drug test positive performed during screening or baseline for any of the following substances:

   1. benzodiazepines,
   2. cocaine,
   3. opioids,
   4. amphetamines,
   5. methamphetamine,
   6. buprenorphine,
   7. methadone,
   8. barbiturates,
   9. oxycodone,
   10. and/or MDMA. Note: Testing for THC was included in the urine drug test; however, subjects who tested positive for THC were still eligible to participate in the study unless they had moderate or greater severity for cannabis use disorder as indicated by DSM-5 criteria. The results for THC were recorded for information only. If positive for opioids or oxycodone but recent opiate use for acute pain was reported by the subject, then the subject could be included at the discretion of the investigator.
3. VAS craving rating ("How strong is your craving to drink alcohol") during first presentation of alcohol cue <5 during the screening cue reactivity session.
4. Have been hospitalized for alcohol intoxication delirium, alcohol withdrawal delirium, alcohol-induced persisting dementia or amnestic disorder, or have had an alcohol withdrawal seizure, alcohol-induced psychotic disorder with a primary diagnosis of AUD or a history of any seizure disorder.
5. Have participated in any behavioral and/or pharmacological intervention research study for the treatment of alcoholism where the last intervention was within 3 years prior to signing the informed consent.
6. Be mandated by the court to obtain treatment for alcohol-dependence, or has probation or parole requirements that might interfere with study participation.
7. Be anyone who in the opinion of the investigator could not be safely withdrawn from alcohol without medical detoxification.
8. Have undergone medical detoxification (e.g., reports using a benzodiazepine) during the screening phase (prior to randomization).
9. Have been treated with a pharmacotherapy for alcohol use disorder within 6 months prior to randomization.
10. Have any of the following, based on DSM-5 criteria as assessed using theMINI:

    1. Current or lifetime diagnosis of psychotic disorders,
    2. Current bipolar disorder,
    3. Current major depressive episode,
    4. Current (past 3 months) eating disorder (anorexia or bulimia), or
    5. Within past year diagnosis of panic disorder with or without agoraphobia. Note: Subjects diagnosed with psychiatric disorders not specifically excluded above could be included at the discretion of the PI as long as the concurrent treatment for the comorbid psychiatric condition does not compromise the study integrity by virtue of its type, duration, or intensity.
11. Have any of the following:

    1. attempted suicide past year,
    2. current (past year) suicide behavior disorder in accordance with DSM-5 criteria as assessed using the MINI (see note below about assessment of subjects diagnosed at low risk),
    3. current (since screening MINI) suicidality risk as indicated during the conduct of the C-SSRS with concurrence after a study physician's evaluation if the response to C-SSRS questions 1 or 2 is "yes"). Note: The MINI suicidality module rates scores of 1 to 8 as a diagnosis of low risk of suicidality. As the MINI questions that could result in a low risk score are considered inadequate to fully determine the potential suicidal risk of an individual (e.g., "Feel hopeless" and "Think that you would be better off dead or wish you were dead?" responses of "yes" dictates a score of 1 for each question), any subject who scores in the low risk category should be evaluated further by a study physician who should document whether the subject is appropriate for study inclusion based on his/her clinical judgment of the potential suicide risk of the subject. Likewise, if the subject responded "yes" to either the first 2 questions on the screening C-SSRS performed on the day of randomization as a final eligibility check, the subject should also have been evaluated by a study physician for current suicidality risk, who should document the subject's suitability for study inclusion.
12. Have moderate or serious dementia as assessed by clinical exam.
13. Be pregnant or breast-feeding or have plans to become pregnant at any time during the study or within 7 days after the last dose of IP.
14. Have clinically significant abnormal laboratory values, including elevation of liver enzymes (AST or ALT > 2.5 x upper limit of normal or total bilirubin > 1.5 x the upper limit of normal).
15. Have abnormal calculated creatinine clearance defined as < 80 mL/minute for subjects ≤ 55 years of age and < 65 mL/minute for subjects > 55 years of age.
16. Have a serious or unstable medical illness or any potentially life-threatening or progressive medical condition other than addiction that may compromise subject safety or study conduct.
17. Be currently undergoing psychotherapy by a licensed therapist or psychiatrist for alcohol problems. NOTE: Current psychotherapy was to be considered on a case-by-case basis. Psychotherapy for a disorder that could be related to the subject's use of alcohol should be exclusionary. However, shorter term focused behavioral therapy for defined problems for non-alcohol related problems could be acceptable.
18. Have data suggesting cirrhosis of the liver (albumin < 3.2 g/dL, or ascites by physical exam).
19. Have been previously treated with ANS-6637 for any reason.
20. Have had gastric bypass surgery.
21. Have had a severe reaction to disulfiram while drinking alcohol requiring medical attention.
22. Have a history of atherosclerotic cardiovascular disease including angina pectoris, myocardial infarction, stroke, transient ischemic attack, peripheral vascular disease or revascularization procedures or clinically significant ECG indicative of cardiovascular disease. Note: medically controlled hypertension is not exclusionary.
23. History of syncope, palpitations, or unexplained dizziness at screening.
24. Had a prior history of any severe adverse reactions to ethanol [e.g., flushing (noticeable redness of the neck or throat) and/or increased heart rate (subject reports sensation of increased heart rate or palpitations) after drinking alcohol].
25. Report heavy drinking of alcohol within 2 days on TLFB prior to screening and have a negative result on EtG urine test.
26. Have Parkinson's Disease or a family history of Parkinson's Disease.
27. Have restless legs syndrome and receiving dopamine agonist treatment.
28. Have attention-deficit disorder and receiving dopamine stimulant treatment.
29. Are taking a prohibited medication.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2019-10-08 (Actual); Primary Completion 2020-05-22 (Actual); Study Completion 2020-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raye Litten, PhD, Study Director — National Institute on Alcohol Abuse and Alcoholism (NIAAA)
Locations (3):
- United States (3):
  - Yale, New Haven, Connecticut
  - Brown University, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No
The data will be shared under a clinical trials agreement with Amygdala Neurosciences.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between October 8, 2019 and May 22, 2020. Participant recruitment methods at each site will be based on their local population; however, standard tactics will be used (including but not limited to: flyers, social media, newspaper advertisements, radio advertisements, and television advertisements).
Pre-assignment Details: n=132 participants were assessed for eligibility. n=89 were excluded prior to randomization for the following reasons: Drinking entry criteria (25%) Screening Cue VAS Score (16%) Vital signs (15%) Positive urine drug test (9%) Other (36%)
Period: Overall Study
Arm/Group | ANS-6637 - 200mg | ANS-6637 - 600mg | Matched Placebo
Started | 15 | 13 | 15
Completed | 14 | 10 | 15
Not Completed | 1 | 3 | 0

BASELINE CHARACTERISTICS:
Population: Sample sizes are based on the modified intention-to-treat (mITT) analysis set, defined as subjects randomized to participate in the study that took at least one dose of IP and had a non-missing VAS craving primary endpoint.
Groups:
- Total: Total of all reporting groups
Arm/Group | ANS-6637 - 200mg | ANS-6637 - 600mg | Matched Placebo | Total
Number analyzed (Participants) | 14 | 10 | 15 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.4 (13.3) | 47.3 (10.1) | 49.8 (12.8) | 46.9 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 2 | 4 | 13
  Male | 7 | 8 | 11 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 2
  Not Hispanic or Latino | 13 | 10 | 14 | 37
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 12 | 10 | 14 | 36
  More than one race | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 10 | 15 | 39
Drinks per Week (28 days before randomization) [Mean (Standard Deviation); unit: standard drinking units (SDUs)] — This is a derived measure of alcohol consumption obtained using a timeline follow-back methodology. A standard drink contains approximately 0.6 fluid ounces (oz) of pure alcohol.
  standard drinking units (SDUs) | 61.2 (20.1) | 46.9 (15.5) | 64.1 (29.8) | 56.6 (24.0)

OUTCOME MEASURES:

1. Primary Outcome: Craving - "How Strong is Your Craving to Drink Alcohol" Visual Analog Scale (VAS) Item
Description: The primary efficacy endpoint is the change in the "strength" of alcohol craving Visual Analog Scale (VAS) score for the question, "How strong is your craving to drink alcohol," in response to an alcohol cue at Week 2 - after one week of investigational product treatment. The VAS has a minimum=0 and maximum=20 with higher values indicative of greater craving for alcohol (a worse outcome).
Time Frame: Week 2
Population: The analysis population is based on the modified intention-to-treat (mITT) analysis set, defined as subjects randomized to participate in the study that took at least one dose of IP and had a non-missing VAS craving primary endpoint.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | ANS-6637 - 200mg | ANS-6637 - 600mg | Matched Placebo
Number analyzed (Participants) | 14 | 10 | 15
score on a scale | 3.91 (1.30) | 6.91 (13.0) | 7.27 (1.25)

2. Secondary Outcome: Number of Subjects With no Heavy Drinking Days
Description: Number of subjects that have no heavy drinking days during the last 4 weeks of treatment. A "heavy drinking day" is 4 or more drinks per drinking day for women and 5 or more drinks per drinking day for men.
Time Frame: Last 4 weeks of treatment, from Week 2 to Week 5
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | ANS-6637 - 200mg | ANS-6637 - 600mg | Matched Placebo
Number analyzed (Participants) | 14 | 10 | 15
Participants | 0 | 2 | 3

3. Secondary Outcome: Number of Subjects Abstinent From Alcohol
Description: Number of subjects that have not drank alcohol during the last 4 weeks of treatment.
Time Frame: Last 4 weeks of treatment, from Week 2 to Week 5
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | ANS-6637 - 200mg | ANS-6637 - 600mg | Matched Placebo
Number analyzed (Participants) | 14 | 10 | 15
Participants | 0 | 1 | 2

4. Secondary Outcome: WHO 1-level Decrease in Alcohol Consumption
Description: The number of subjects experiencing at least a 1-level decrease in World Health Organization (WHO) levels of alcohol consumption from the level at baseline (the period including the 28 days before screening) to the level during the last 4 weeks of treatment.
  The WHO levels of average alcohol consumption per day are as follows:
  Males Females Low Risk 1 to 40g 1 to 20g Medium Risk 41 to 60g 21 to 40g High Risk 61 to 100g 41 to 60g Very High Risk 101+g 61+g where 14g = 1 SDU (WHO-2000). In computing the WHO alcohol consumption level, average drinks per day were used, computed as the sum of all drinks in the 28 day period divided by the number of days with non-missing drinking data in that period. Abstinent subjects were included in a separate "Abstinent" category.
Time Frame: Last 4 weeks of treatment, from Week 2 to Week 5
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | ANS-6637 - 200mg | ANS-6637 - 600mg | Matched Placebo
Number analyzed (Participants) | 14 | 10 | 15
Participants | 12 | 10 | 10

5. Secondary Outcome: WHO 2-level Decrease in Alcohol Consumption
Description: The number of subjects experiencing at least a 2-level decrease in World Health Organization (WHO) levels of alcohol consumption from the level at baseline (the period including the 28 days before screening) to the level during the last 4 weeks of treatment.
  The WHO levels of average alcohol consumption per day are as follows:
  Males Females Low Risk 1 to 40g 1 to 20g Medium Risk 41 to 60g 21 to 40g High Risk 61 to 100g 41 to 60g Very High Risk 101+g 61+g where 14g = 1 SDU (WHO-2000). In computing the WHO alcohol consumption level, average drinks per day were used, computed as the sum of all drinks in the 28 day period divided by the number of days with non-missing drinking data in that period. Abstinent subjects were included in a separate "Abstinent" category.
Time Frame: Last 4 weeks of treatment, from Week 2 to Week 5
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | ANS-6637 - 200mg | ANS-6637 - 600mg | Matched Placebo
Number analyzed (Participants) | 14 | 10 | 15
Participants | 6 | 6 | 5

6. Secondary Outcome: Percentage of Days Abstinent
Description: The percentage of days abstinent from drinking alcohol
Time Frame: Last 4 weeks of treatment, from Week 2 to Week 5
Population: mITT
Measure: Mean (95% Confidence Interval); unit: percentage of days abstinent
Arm/Group | ANS-6637 - 200mg | ANS-6637 - 600mg | Matched Placebo
Number analyzed (Participants) | 14 | 10 | 15
percentage of days abstinent | 32.3 [19.3 to 53.2] | 51.3 [30.8 to 71.8] | 38.1 [21.4 to 54.8]

7. Secondary Outcome: Percentage of Heavy Drinking Days
Description: Percentage of heavy drinking days where a heavy drinking day is 4 or more drinks on a day for women or 5 or more drinks on a day for men.
Time Frame: Last 4 weeks of treatment, from Week 2 to Week 5
Population: mITT
Measure: Mean (95% Confidence Interval); unit: percentage of heavy drinking days
Arm/Group | ANS-6637 - 200mg | ANS-6637 - 600mg | Matched Placebo
Number analyzed (Participants) | 14 | 10 | 15
percentage of heavy drinking days | 37.0 [20.5 to 53.5] | 26.5 [6.0 to 47.1] | 40.8 [25.0 to 56.7]

8. Secondary Outcome: Percentage of Very Heavy Drinking Days
Description: Percentage of very heavy drinking days where a very heavy drinking day is defined as 8 or more drinks on a day for women and 10 or more drinks on a day for men.
Time Frame: Last 4 weeks of treatment, from Week 2 to Week 5
Population: mITT
Measure: Mean (95% Confidence Interval); unit: percentage of very heavy drinking days
Arm/Group | ANS-6637 - 200mg | ANS-6637 - 600mg | Matched Placebo
Number analyzed (Participants) | 14 | 10 | 15
percentage of very heavy drinking days | 8.0 [-0.2 to 16.2] | 3.8 [-6.2 to 13.7] | 9.1 [1.2 to 17.0]

9. Secondary Outcome: Drinks Per Week
Description: The number of drinks consumed per week
Time Frame: Last 4 weeks of treatment, from Week 2 to Week 5
Population: mITT
Measure: Mean (95% Confidence Interval); unit: standard drinking units (SDUs)
Arm/Group | ANS-6637 - 200mg | ANS-6637 - 600mg | Matched Placebo
Number analyzed (Participants) | 14 | 10 | 15
standard drinking units (SDUs) | 24.3 [14.6 to 34.0] | 19.0 [6.8 to 31.1] | 27.2 [17.7 to 36.7]

10. Secondary Outcome: Drinks Per Drinking Day
Description: The number of drinks consumed on days where participants drank
Time Frame: Last 4 weeks of treatment, from Week 2 to Week 5
Population: mITT
Measure: Mean (95% Confidence Interval); unit: standard drinking units (SDUs)
Arm/Group | ANS-6637 - 200mg | ANS-6637 - 600mg | Matched Placebo
Number analyzed (Participants) | 14 | 10 | 15
standard drinking units (SDUs) | 5.4 [4.4 to 6.4] | 4.7 [3.3 to 6.1] | 6.1 [5.1 to 7.2]

11. Secondary Outcome: Penn Alcohol Craving Scale (PACS)
Description: The amount of craving; higher numbers indicate more craving. There are 5 items each on a 0 to 6 scale. Items are summed to get to the total craving, resulting in scores having a min=0 and max=30.
Time Frame: Last 4 weeks of treatment, from Week 2 to Week 5
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | ANS-6637 - 200mg | ANS-6637 - 600mg | Matched Placebo
Number analyzed (Participants) | 14 | 10 | 15
score on a scale | 12.0 [9.5 to 14.5] | 11.3 [8.4 to 14.2] | 12.0 [9.6 to 14.3]

12. Secondary Outcome: Pittsburgh Sleep Quality Index (PSQI)
Description: A measure of sleep quality; the PSQI includes a scoring key for calculating a patient's seven subscores, each of which can range from 0 to 3. The subscores are tallied, yielding a "global" score that can range from 0 to 21. A global score of 5 or more indicates poor sleep quality; the higher the score, the worse the quality.
Time Frame: Last 4 weeks of treatment, from Week 2 to Week 5
Population: mITT
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | ANS-6637 - 200mg | ANS-6637 - 600mg | Matched Placebo
Number analyzed (Participants) | 14 | 10 | 15
score on a scale | 6.6 [5.1 to 8.1] | 6.2 [4.6 to 7.9] | 5.0 [3.8 to 6.3]

13. Secondary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS) Alcohol Related Negative Consequences
Description: A measure of alcohol-related negative consequences. There are 7 items scored on a 1 to 7 scale (a higher score indicative greater frequency of negative consequences). The items are summed and converted to a T-score to create a total score. The T-scores range from 0 to 100 (the population mean = 50 and standard deviation = 10). Higher T-scores are indicative of more negative consequences (worse outcome).
Time Frame: Last 4 weeks of treatment, from Week 2 to Week 5
Population: mITT
Measure: Mean (95% Confidence Interval); unit: T-score
Arm/Group | ANS-6637 - 200mg | ANS-6637 - 600mg | Matched Placebo
Number analyzed (Participants) | 14 | 10 | 15
T-score | 47.8 [44.7 to 50.4] | 45.9 [42.3 to 49.6] | 50.7 [50.0 to 53.3]

14. Secondary Outcome: Profile of Mood States (POMS) Total Disturbance
Description: A measure of total mood disturbance. Total mood disturbance is the sum of depression, anger, fatigue, confusion, and tension subscales subtracting the vigor subscale items. The range of possible scores is from -32 to 200 with higher scores indicating greater mood disturbance.
Time Frame: Last 4 weeks of treatment, from Week 2 to Week 5
Population: mITT
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | ANS-6637 - 200mg | ANS-6637 - 600mg | Matched Placebo
Number analyzed (Participants) | 14 | 10 | 15
score on a scale | -2.0 [-12.9 to 8.9] | 3.9 [-7.8 to 15.7] | 9.1 [-0.4 to 18.7]

15. Secondary Outcome: Craving - "Having a Drink Would Making Things Just Perfect" Visual Analog Scale (VAS) Item
Description: This secondary efficacy endpoint is the change in the Visual Analog Scale (VAS) score for the question, "Having a drink would make things just perfect," in response to an alcohol cue at Week 2 - after one week of investigational product treatment. The VAS has a minimum=0 and maximum=20 with higher values indicative of greater craving for alcohol (a worse outcome).
Time Frame: Week 2
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | ANS-6637 - 200mg | ANS-6637 - 600mg | Matched Placebo
Number analyzed (Participants) | 14 | 10 | 15
score on a scale | 3.72 (1.43) | 5.23 (3.72) | 6.38 (1.40)

16. Secondary Outcome: Craving - "If I Could Drink Alcohol Now, I Would Drink it" Visual Analog Scale (VAS) Item
Description: This secondary efficacy endpoint is the change in the Visual Analog Scale (VAS) score for the question, "If I could drink alcohol now, I would drink it," in response to an alcohol cue at Week 2 - after one week of investigational product treatment. The VAS has a minimum=0 and maximum=20 with higher values indicative of greater craving for alcohol (a worse outcome).
Time Frame: Week 2
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | ANS-6637 - 200mg | ANS-6637 - 600mg | Matched Placebo
Number analyzed (Participants) | 14 | 10 | 15
score on a scale | 5.67 (1.65) | 8.41 (2.05) | 6.69 (1.63)

17. Secondary Outcome: Craving - "It Would be Hard to Turn Down a Drink Right Now" Visual Analog Scale (VAS) Item
Description: This secondary efficacy endpoint is the change in the Visual Analog Scale (VAS) score for the question, "It would be hard to turn down a drink right now," in response to an alcohol cue at Week 2 - after one week of investigational product treatment. The VAS has a minimum=0 and maximum=20 with higher values indicative of greater craving for alcohol (a worse outcome).
Time Frame: Week 2
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | ANS-6637 - 200mg | ANS-6637 - 600mg | Matched Placebo
Number analyzed (Participants) | 14 | 10 | 15
score on a scale | 3.37 (1.42) | 7.46 (1.74) | 6.82 (1.38)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during the entire 8 weeks study period (6 weeks of treatment + 2 weeks follow-up after treatment).
Arm/Group | ANS-6637 - 200mg | ANS-6637 - 600mg | Matched Placebo
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/13 | 0/15
Serious Adverse Events (participants affected / at risk) | 2/15 | 1/13 | 0/15
Other Adverse Events (participants affected / at risk) | 15/15 | 13/13 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ANS-6637 - 200mg (N=15) | ANS-6637 - 600mg (N=13) | Matched Placebo (N=15)
Alcohol Rehabilitation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Drug-Induced Liver Injury (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Alanine-Aminotransferase Increased (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ANS-6637 - 200mg (N=15) | ANS-6637 - 600mg (N=13) | Matched Placebo (N=15)
BRADYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
PALPITATIONS (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
SINUS BRADYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2)
EAR DISCOMFORT (Ear and labyrinth disorders) | 1 (3) | 0 (0) | 0 (0)
PHOTOPSIA (Eye disorders) | 1 (3) | 0 (0) | 0 (0)
VISION BLURRED (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
DRY MOUTH (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
DYSPEPSIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 2 (2) | 5 (6) | 1 (2)
SWOLLEN TONGUE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
TONGUE DISCOMFORT (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
TOOTHACHE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
VOMITING (Gastrointestinal disorders) | 1 (2) | 3 (3) | 0 (0)
ASTHENIA (General disorders) | 1 (1) | 0 (0) | 0 (0)
CHEST PAIN (General disorders) | 1 (2) | 0 (0) | 1 (1)
CHILLS (General disorders) | 1 (1) | 0 (0) | 0 (0)
FATIGUE (General disorders) | 3 (4) | 1 (1) | 3 (3)
FEELING ABNORMAL (General disorders) | 0 (0) | 0 (0) | 1 (1)
FEELING COLD (General disorders) | 1 (1) | 0 (0) | 0 (0)
FEELING HOT (General disorders) | 1 (1) | 1 (2) | 3 (5)
INFLUENZA LIKE ILLNESS (General disorders) | 1 (1) | 0 (0) | 1 (1)
PYREXIA (General disorders) | 1 (1) | 0 (0) | 0 (0)
BRONCHITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
FUNGAL INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 1 (1) | 2 (2) | 1 (1)
ALCOHOL POISONING (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
CONCUSSION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
FACIAL BONES FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
LIMB INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 3 (6) | 4 (5) | 4 (4)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 4 (7) | 4 (4) | 3 (3)
BLOOD ALBUMIN DECREASED (Investigations) | 1 (1) | 0 (0) | 0 (0)
BLOOD ALKALINE PHOSPHATASE DECREASED (Investigations) | 1 (1) | 0 (0) | 0 (0)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0)
BLOOD BILIRUBIN INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0)
BLOOD CREATININE DECREASED (Investigations) | 2 (3) | 1 (1) | 2 (3)
BLOOD PRESSURE DIASTOLIC INCREASED (Investigations) | 2 (2) | 5 (9) | 5 (5)
BLOOD PRESSURE INCREASED (Investigations) | 1 (1) | 0 (0) | 1 (1)
BLOOD PRESSURE SYSTOLIC INCREASED (Investigations) | 5 (6) | 3 (3) | 3 (3)
BLOOD THYROID STIMULATING HORMONE DECREASED (Investigations) | 4 (5) | 6 (8) | 1 (1)
EOSINOPHIL COUNT DECREASED (Investigations) | 0 (0) | 1 (1) | 0 (0)
EOSINOPHIL COUNT INCREASED (Investigations) | 1 (1) | 0 (0) | 2 (2)
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 2 (4) | 1 (1) | 0 (0)
GLUCOSE URINE PRESENT (Investigations) | 1 (1) | 0 (0) | 0 (0)
HAEMATOCRIT DECREASED (Investigations) | 3 (3) | 3 (3) | 2 (2)
HEART RATE INCREASED (Investigations) | 9 (12) | 9 (11) | 1 (2)
LYMPHOCYTE COUNT DECREASED (Investigations) | 1 (1) | 0 (0) | 1 (1)
LYMPHOCYTE COUNT INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0)
MONOCYTE COUNT INCREASED (Investigations) | 2 (2) | 2 (2) | 0 (0)
NEUTROPHIL COUNT DECREASED (Investigations) | 0 (0) | 1 (1) | 2 (2)
NEUTROPHIL COUNT INCREASED (Investigations) | 1 (1) | 0 (0) | 1 (1)
PLATELET COUNT DECREASED (Investigations) | 0 (0) | 0 (0) | 1 (1)
PLATELET COUNT INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1)
RED BLOOD CELL COUNT DECREASED (Investigations) | 5 (5) | 2 (2) | 4 (4)
THYROXINE DECREASED (Investigations) | 0 (0) | 0 (0) | 2 (2)
THYROXINE FREE DECREASED (Investigations) | 0 (0) | 0 (0) | 1 (1)
THYROXINE FREE INCREASED (Investigations) | 3 (3) | 6 (7) | 0 (0)
THYROXINE INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0)
TRI-IODOTHYRONINE DECREASED (Investigations) | 0 (0) | 0 (0) | 1 (1)
TRI-IODOTHYRONINE INCREASED (Investigations) | 5 (5) | 5 (6) | 0 (0)
VITAMIN D DECREASED (Investigations) | 0 (0) | 1 (1) | 0 (0)
WEIGHT INCREASED (Investigations) | 0 (0) | 2 (3) | 0 (0)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 2 (2) | 1 (1) | 0 (0)
WHITE BLOOD CELL COUNT INCREASED (Investigations) | 3 (3) | 0 (0) | 1 (1)
ALCOHOL INTOLERANCE (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 2 (2) | 4 (4) | 3 (3)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
FOOD CRAVING (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
INCREASED APPETITE (Metabolism and nutrition disorders) | 5 (5) | 4 (5) | 6 (6)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
DIZZINESS (Nervous system disorders) | 2 (2) | 1 (1) | 1 (2)
HEADACHE (Nervous system disorders) | 4 (5) | 3 (4) | 6 (9)
HYPOAESTHESIA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
PARAESTHESIA (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2)
RESTLESS LEGS SYNDROME (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
TREMOR (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
ALCOHOL WITHDRAWAL SYNDROME (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
ALCOHOLIC HANGOVER (Psychiatric disorders) | 1 (1) | 0 (0) | 2 (2)
ALCOHOLISM (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
ANXIETY (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
DRUG ABUSE (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
EMOTIONAL DISORDER (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
INSOMNIA (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
IRRITABILITY (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
CHROMATURIA (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
POLLAKIURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (4)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
PRURITUS (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
DENTAL OPERATION (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
FLUSHING (Vascular disorders) | 10 (10) | 11 (11) | 2 (2)
HOT FLUSH (Vascular disorders) | 2 (2) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PIs may only publish on study results after the main results are published.

DOCUMENTS (3):
  • Study Protocol (2020-03-27): https://cdn.clinicaltrials.gov/large-docs/09/NCT03970109/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-16): https://cdn.clinicaltrials.gov/large-docs/09/NCT03970109/SAP_001.pdf
  • Informed Consent Form (2020-05-26): https://cdn.clinicaltrials.gov/large-docs/09/NCT03970109/ICF_002.pdf